CLINICAL TRIAL: NCT01752543
Title: Effects on Exercise Hemodynamics of Vasopressin Blockade by Conivaptan Infusion in Heart Failure Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Finn Gustafsson (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Finn Gustafsson, Staff Cardiologist, MD, Phd, DMSci, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: H-3-2012-139
Record Dates: First submitted 2012-12-12; First posted 2012-12-19 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Heart Failure
Keywords: Vasopressin; Exercise capacity; Conivaptan
MeSH Terms: conditions — Heart Failure; Diabetes Insipidus | interventions — conivaptan; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conivaptan (Active Comparator): 10 patients will be randomized to conivaptan treatment
  Interventions: Drug: Conivaptan
- Dextrose (Placebo Comparator): 10 patients will receive placebo treatment (dextrose)
  Interventions: Drug: Placebo (Dextrose)

INTERVENTIONS:
Drug: Conivaptan — Conivaptan treatment: 20 mg bolus followed by infusion of 2 mg/hour
  Other Names: Vaprisol
  Arms: Conivaptan
Drug: Placebo (Dextrose) — Placebo treatment: 20 mg bolus followed by infusion of 2 mg/hour
  Other Names: 5 % dextrose
  Arms: Dextrose

SUMMARY:
The purpose of the present study is to evaluate the effects of a blockade of the vasopressin system and central hemodynamic system in heart failure (HF) patients during physical exercise. The significance of the vasopressin system during physical exercise is unclear. If vasopressin is a significant regulator of exercise hemodynamics in HF, strategies to intervene against activation of the V1A-receptor might be expected to improve HF symptoms and possibly outcome.

The potential effects of the central hemodynamic system will be evaluated with a Swan-Ganz catheter. Echocardiography will be performed at rest and during submaximal working capacity before and during the infusion of a vasopressin receptor antagonist (conivaptan) or placebo. Cardiac output will be measured by thermodilution. The exercise test will be performed at 50 % of VO2 max and hemodynamic and echocardiographic measurements will be collected. The exercise test will be performed on a supine multistage bicycle.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Left ventricular ejection fraction (LVEF) < 45 % on the baseline echocardiography.
* Treatment with beta-blockers and angiotensin-converting-enzyme (ACE) inhibitors for at least 1 month as tolerated
* New York Heart Association (NYHA) Functional Class II-III
* Given informed consent
* Women, who have not yet entered menopause (defined as no menstrual bleeding in the last 12 months), will provide a negative urine HCG before entering the study

Exclusion Criteria:

* Signs of symptomatic or ongoing myocardial ischemia
* Known non-revascularized coronary disease
* Presence of hypovolemic hyponatremia (P-Na+ <130 mmol/l and clinical signs of volume depletion or dehydration as judged by investigator).
* Hypernatraemia (P-Na+) > 145 mmol/L
* Chronic obstructive pulmonary disease (FEV1/FVC < 70 % and/or 30 % > FEV1 < 50 %)
* Supine systolic blood pressure < 85 mmHg
* Significant orthostatic hypotension
* Standing blood pressure < 80 mmHg or a blood pressure drop > 20 mmHg when changing from a supine to a standing position
* Uncontrolled hypertension evaluated by the investigator
* Uncontrolled cardiac arrhythmias evaluated by the investigator
* Untreated serious hypothyroidism
* Adrenal insufficiency
* Poor echocardiographic window
* Inability to perform exercise testing
* Permanent atrial fibrillation or atrial fluttering
* Planned coronary by-pass surgery
* Moderate hepatic impairment (ALAT/ASAT > 3 UNL)
* Presence of other diseases affecting treatment with conivaptan or the evaluation of safety as evaluated by the investigator
* Severely decreased kidney function (eGFR < 20 mL/min)
* Serum K+< 3.5 or > 5.5 mmol/L
* Known conivaptan intolerability
* Corn allergy
* Dextrose Allergy
* Treatment with potent CYP3A-inhibitors (ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir)
* Treatment with arginine vasopressin, oxytocin, desmopressin and other medications for the treatment of hyponatremia (lithium salts, urea and demeclocycline)
* Warfarin treatment
* Presence of infection or active bleeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The joint endpoint of change in pulmonary capillary wedge pressure (PCWP) and cardiac output (CO) at the submaximal exercise intensity of 50 % of the maximal exercise capacity | 1 day

SECONDARY OUTCOMES:
Cardiac index (CI) during submaximal exercise from rest to submaximal exercise | 1 day
Pulmonary and systemic vascular resistance from rest to submaximal exercise | 1 day
Left ventricular end diastolic diameter during exercise from rest to submaximal exercise | 1 day
The change in mean pulmonary artery pressure (mPAP) from rest to submaximal exercise | 1 day
The change in BNP, MR-ANP and copeptin from rest to submaximal exercise | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Louise Balling, MD, Principal Investigator — Rigshospitalet, Denmark; Finn Gustafsson, MD, PhD, DMSci, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Cardiology, Copenhagen University Hospital, Rigshospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Balling L, Thomsen JH, Wolsk E, Hassager C, Boesgaard S, Goldsmith SR, Gustafsson F. Hemodynamic effects of short-term infusion of a vasopressin V1A/V2 receptor antagonist conivaptan in patients withchronic heart failure during submaximal exercise. Am Heart J. 2018 Sep;203:101-104. doi: 10.1016/j.ahj.2018.05.015. Epub 2018 Jun 14. No abstract available. PMID 30057012